CLINICAL TRIAL: NCT01033669
Title: A Randomized Cross-Over Study Investigating The Inhalation Profiles Of Four Dry Powder Inhalation Devices In Subjects With Asthma And Chronic Obstructive Pulmonary Disease.
Brief Title: Assessment Of The Inhalation Profiles Of Four Dry Powder Inhalers In Patients With Variable Degrees Of Lung Obstruction
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A9011071
Record Dates: First submitted 2009-09-24; First posted 2009-12-16 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Asthma; Pulmonary Disease, Chronic Obstructive
Keywords: Inhalation profiles; asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dry Powder Inhalers
  Interventions: Device: CRC-749; Device: Diskus; Device: Twisthaler; Device: Miat Monohaler

INTERVENTIONS:
Device: CRC-749 — There is no drug being used. This is a device.
Device: Diskus — There is no drug being used. This is a device.
Device: Twisthaler — There is no drug being used. This is a device.
Device: Miat Monohaler — There is no drug being used. This is a device.

SUMMARY:
Assessment of the inhalation profiles of four dry powder inhalers in patients with variable degrees of lung obstruction

DETAILED DESCRIPTION:
Randomized to device sequence

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a physician documented history or diagnosis of asthma for at least 6 months
* Reversibility, defined as an increase in FEV1 at the Screening visit of greater than or equal to 12% and 200 mL
* Subjects with a physician documented history or diagnosis of mild or severe Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* Female subjects who are pregnant
* Subjects who have a history of life-threatening asthma/COPD or who have experienced two or more exacerbations requiring hospitalization in the 12 months prior to screening
* Evidence of lower respiratory tract infection
* Subjects diagnosed with pulmonary fibrosis, bronchiectasis, pneumoconiosis, sarcoidosis or tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma and COPD patients
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Peak Inspiratory Flow Rate | Day 3-10

SECONDARY OUTCOMES:
Pressure Slope | Day 3-10
Peak Pressure Drop | Day 3-10
Time to Peak Pressure Drop | Day 3-10
Inhaled Volume | Day 3-10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Berlin, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011071&StudyName=Assessment%20Of%20The%20Inhalation%20Profiles%20Of%20Four%20Dry%20Powder%20Inhalers%20In%20Patients%20With%20Variable%20Degrees%20Of%20Lung%20Obstruction